CLINICAL TRIAL: NCT02444715
Title: Study on Improved Prevention Methods for Cerebro-cardiovascular Diseases Based on a Computer-aided Prevention System
Brief Title: Computer-Aided Prevention System
Acronym: CAPSYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lübomira Spassova (Other)
Collaborators: Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor-Investigator, Lübomira Spassova, Dr.-Ing., Luxembourg Institute of Science and Technology
Organization: Luxembourg Institute of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAPSYS-201205/08-1
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Cerebrovascular Diseases; Stroke; Cardiovascular Diseases; CVD Risk Factors
Keywords: Lifestyle coaching; Phone-based system; CVD prevention; Patient-centered decision support
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke; Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (SC) (Active Comparator)
  Interventions: Behavioral: Standard care
- Interventional care (IC) (Experimental)
  Interventions: Behavioral: CAPSYS

INTERVENTIONS:
Behavioral: Standard care — Participants receive only the usual care including blood analyses, blood pressure controls and individual advice on healthy lifestyle during the outpatient treatment given by the neurologist, by the general practitioner and by other physicians.
  Arms: Standard care (SC)
Behavioral: CAPSYS — In addition to the usual care, patients are asked to call the CAPSYS system twice a week.
  Arms: Interventional care (IC)

SUMMARY:
Stroke is one of the most frequent and life-threatening diseases in Europe. About four stroke events occur per day in Luxembourg alone, and about 30% of these patients are affected by recurrent stroke within the following five years. Thus, new methods of primary and secondary prevention are needed to better control lifestyle-related risk factors.

The development and maintenance of a healthy lifestyle (smoking cessation, healthy nutrition, moderate physical exercises etc.) is a major objective concerning the primary and secondary prevention of cerebro- and cardiovascular diseases. CAPSYS is a computer-based lifestyle coaching system developed by researchers from the Public Research Centre (CRP) Henri Tudor in Luxembourg in collaboration with neurologists from the Centre Hospitalier de Luxembourg (CHL), which aims at supporting patients in performing appropriate behavior changes in order to minimize their individual risk factors. Patients can access CAPSYS by dialing a local-rate telephone number and answer to a set of previously known questions concerning their current nutrition, physical activity, blood pressure, smoking etc. In an interactive voice response approach, questions are issued by the system in natural language using text-to-speech, and the patient can provide the required values using the phone keypad. Based on the gathered values for each patient, the system automatically generates personalized verbal feedback at runtime and presents it to the patient during the phone dialog. Depending on the individual development of the patient's risk factors, the system feedback can contain advice for improvement, praise for healthy behavior and motivation to pursue a certain goal.

The user acceptance and effectiveness of the CAPSYS system is evaluated in a six-month randomized controlled study with participants recruited at CHL's neurology department.

ELIGIBILITY:
Inclusion Criteria:

* At high risk of stroke:

  * Already suffered a stroke or Transient Ischemic Attack (TIA) or
  * At least two risk factors for stroke:

    * High blood pressure
    * Overweight
    * Low physical activity
    * Smoking
    * Unhealthy diet

Exclusion Criteria:

* Inability to fill out or to understand the informed consent
* No signed informed consent
* Dementia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lübomira Spassova, Dr.-Ing., Study Chair — Luxembourg Institute of Science and Technology; Debora Vittore, Study Chair — Centre Hospitalier de Luxembourg (CHL); Dirk W Droste, Prof. Dr., Principal Investigator — Centre Hospitalier de Luxembourg (CHL); Norbert Rösch, Prof. Dr., Study Director — University of Applied Sciences Kaiserslautern

REFERENCES:
- [Background] Spassova L, Vittore D, Droste D, Rosch N. Automated lifestyle coaching for cerebro-cardiovascular disease prevention. Stud Health Technol Inform. 2013;190:234-6. PMID 23823433
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Spassova L, Vittore D, Droste DW, Rosch N. Randomised controlled trial to evaluate the efficacy and usability of a computerised phone-based lifestyle coaching system for primary and secondary prevention of stroke. BMC Neurol. 2016 Feb 9;16:22. doi: 10.1186/s12883-016-0540-4. PMID 26861865

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Started | 46 | 48
Completed | 36 | 32
Not Completed | 10 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care (SC) | Interventional Care (IC) | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (12.1) | 60.7 (11.3) | 60.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 29 | 34 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Time Frame: baseline and 6 months
Population: Blood pressure data is missing for 4 of the 36 SC and 4 of the 32 IC participants who provided final questionnaires.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 32 | 28
mmHg | 0.19 (21.34) | -9 (21.37)
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.96, t-test, 2 sided
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

2. Primary Outcome: Change in HDL Level
Time Frame: baseline and 6 months
Population: For participants who did not provide final questionnaires, data was retrieved from medical records. HDL data is missing for 5 of the 46 SC and 11 of the 48 IC participants who started the study.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 41 | 37
mg/dl | 1 [-5 to 7] | -2 [-7 to 4]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.44, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in LDL Level
Time Frame: baseline and 6 months
Population: For participants who did not provide final questionnaires, data was retrieved from medical records. LDL data is missing for 5 of the 46 SC and 11 of the 48 IC participants who started the study.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 41 | 37
mg/dl | -1 [-17 to 10] | -6 [-16 to 3]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Triglyceride Level
Time Frame: baseline and 6 months
Population: For participants who did not provide final questionnaires, data was retrieved from medical records. Triglyceride data is missing for 16 of the 46 SC and 16 of the 48 IC participants who started the study.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 30 | 32
mg/dl | -1 [-33.25 to 18] | -11 [-37.5 to 10.25]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Change in HbA1c Level
Time Frame: baseline and 6 months
Population: For participants who did not provide final questionnaires, data was retrieved from medical records. HbA1c data is missing for 21 of the 46 SC and 21 of the 48 IC participants who started the study.
Measure: Median (Inter-Quartile Range); unit: percent HbA1c
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 25 | 27
percent HbA1c | -0.1 [-0.2 to 0.2] | -0.1 [-0.2 to 0]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Change in Glycaemia Level
Time Frame: baseline and 6 months
Population: For participants who did not provide final questionnaires, data was retrieved from medical records. Glycaemia data is missing for 6 of the 46 SC and 13 of the 48 IC participants who started the study.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 40 | 35
mg/dl | -0.5 [-8.25 to 6] | -2 [-7.5 to 2.5]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Change in BMI Value
Time Frame: baseline and 6 months
Population: For participants who did not provide final questionnaires, data was retrieved from medical records. Weight data is missing for 9 of the 46 SC and 15 of the 48 IC participants who started the study.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 37 | 33
kg/m^2 | 0.05 (1.61) | -0.26 (1.3)
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.9, t-test, 2 sided
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

8. Secondary Outcome: Change in Fruits and Vegetables Consumption
Description: Self-reported weekly portions of fruits and vegetables consumption
  (During the recruiting interview, participants were instructed in estimating the size of a portion of fruits or vegetables and they were provided an information booklet on this topic.)
Time Frame: baseline and 6 months
Population: Data on fruits and vegetables consumption was retrieved from final questionnaires. Hence, food consumption data is missing for the 10 SC and 16 IC participants who did not provide final questionnaires.
Measure: Median (Inter-Quartile Range); unit: portions
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 36 | 32
portions | 0 [-7 to 7] | 3.5 [-3.25 to 11.75]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.67, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Whole Grain Food Consumption
Description: Self-reported weekly portions of whole grain food consumption
  (During the recruiting interview, participants were instructed in estimating the size of a portion of whole grain food and they were provided an information booklet on this topic.)
Time Frame: baseline and 6 months
Population: Data on whole grain food consumption was retrieved from final questionnaires. Hence, food consumption data is missing for the 10 SC and 16 IC participants who did not provide final questionnaires.
Measure: Median (Inter-Quartile Range); unit: portions
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 36 | 32
portions | 0 [-4 to 3] | 1 [-0.25 to 7]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Sweets Consumption
Description: Self-reported weekly portions of sweets consumption
  (During the recruiting interview, participants were instructed in estimating the size of a portion of sweets and they were provided an information booklet on this topic.)
Time Frame: baseline and 6 months
Population: Data on sweets consumption was retrieved from final questionnaires. Hence, food consumption data is missing for the 10 SC and 16 IC participants who did not provide final questionnaires.
Measure: Median (Inter-Quartile Range); unit: portions
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 36 | 32
portions | 0 [0 to 1] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Duration of Physical Activity
Description: Self-reported weekly duration of physical activity of medium or high intensity
Time Frame: baseline and 6 months
Population: Data on physical activity was retrieved from final questionnaires. Hence, physical activity data is missing for the 10 SC and 16 IC participants who did not provide final questionnaires.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 36 | 32
minutes
  medium intensity | 0 [-60 to 135] | 0 [-60 to 112.5]
  high intensity | 0 [-120 to 15] | 0 [-45 to 30]
Statistical Analysis 1: Comparison: Standard Care (SC); Medium intensity H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); Medium intensity H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard Care (SC); High intensity H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Interventional Care (IC); High intensity H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Quality of Life
Description: The QoL was measured using the standardised EQ-5D-5L instrument provided by the EuroQol Group.
  In this context, the health value was specified by the participants on a subjective scale ranging from 0 ("The worst health you can imagine") to 100 ("The best health you can imagine").
Time Frame: baseline and 6 months
Population: Data on quality of life was retrieved from final questionnaires. Hence, QoL data is missing for the 10 SC and 16 IC participants who did not provide final questionnaires.
Measure: Median (Inter-Quartile Range); unit: units on a scale (health value)
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Number analyzed (Participants) | 36 | 32
units on a scale (health value) | 0 [-6.25 to 10] | 0 [-0.25 to 5]
Statistical Analysis 1: Comparison: Standard Care (SC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interventional Care (IC); H0: no change between baseline and post-intervention; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)

13. Other Pre Specified Outcome: Usability: SUS Score
Description: The usability of the intervention was assessed based on the standardised System Usability Scale (SUS).
  SUS scores were not collected in the SC group because the SC participants were not using CAPSYS and hence were not able to assess its usability.
  The System Usability Scale (SUS) provides a "quick and dirty", reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Originally created by John Brooke in 1986, it allows to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications.
  The total SUS score computed based on the responses provided to each of the 10 items can range from 0 (worst) to 100 (best). Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average.
Time Frame: 6 months
Population: SUS questionnaires are missing, incomplete or invalid for 6 of the 32 IC participants who provided final questionnaires.
Measure: Mean (Standard Deviation); unit: units on a scale (total SUS score)
Arm/Group | Interventional Care (IC)
Number analyzed (Participants) | 26
units on a scale (total SUS score) | 80.1 (16.22)

ADVERSE EVENTS:
Arm/Group | Standard Care (SC) | Interventional Care (IC)
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No